CLINICAL TRIAL: NCT05430997
Title: Hypothermia Risk Prediction Combined With Active Insulation Management in the Burden of Disease Study in Geriatric Surgery: A Multicenter, Randomized, Controlled Study Based on 24 Hospitals in Southwest China
Brief Title: Hypothermia Risk Prediction Combined With Active Insulation Management in Geriatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Min Su, Professor.Min, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BTM-20220608
Record Dates: First submitted 2022-06-14; First posted 2022-06-24 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Hypothermia; Anesthesia; Body Temperature Changes
MeSH Terms: conditions — Hypothermia; Body Temperature Changes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: conventional management (Active Comparator): The ambient temperature of the operating room was set at 23±2 ℃ and the relative humidity was 50% to 60%. Intraoperative infusion fluids, blood products and rinsing fluid were warmed. Patients were given quilts to cover after entering the operating room, and the quilts covered from the neck to both the feet.
  Interventions: Device: cover with a quilt from the neck to both feet
- Group B: Hypothermia Risk Prediction Joint Active Insulation Management (Experimental): In the test group, after the assessment of the "Intraoperative Hypothermia Risk Prediction APP", patients who were "prompted/recommended to use active warming measures" were actively warmed by inflatable warming (IOB Warming Unit (WU505) + Inflatable Warming Blanket) after admission to the room. Warming Unit (WU505) + Warming Blanket (IOB Warming Blanket)) was used for active warming. The air inlet was connected to the air catheter, and the host temperature was set at 38 ℃ with "high" air speed. During the operation, the thermal blanket is covered with non-surgical sterilization area (such as both shoulders, torso, healthy limbs, etc.), and the host temperature is adjusted to 38 ℃ for thermal insulation. The temperature and wind speed were adjusted in time to maintain the oropharyngeal temperature at 36.2℃～37.2℃ by monitoring the body temperature at any time during the operation.
  Interventions: Device: IOB Warming Unit (WU505) + Inflatable Warming Blanket

INTERVENTIONS:
Device: IOB Warming Unit (WU505) + Inflatable Warming Blanket — The inflatable warming method (Inflatable Warming Unit (IOB Warming Unit, WU505) + Inflatable Warming Blanket (IOB Warming Blanket)) is a common clinical warming technique in anesthesiology, which is well tolerated by patients and safe and effective. The anesthesiology department has established standard operating procedures for the above-mentioned non-invasive operations.
  Arms: Group B: Hypothermia Risk Prediction Joint Active Insulation Management
Device: cover with a quilt from the neck to both feet — The patient was covered with a quilt from the neck to both feet after entering the operating room.
  Arms: Group A: conventional management

SUMMARY:
To evaluate the effectiveness and safety of hypothermia risk prediction combined with active warming management to reduce intraoperative hypothermia in elderly patients undergoing elective general anesthesia, improve the quality of anesthesia management, and enhance patients' awareness of the work of anesthesiologists.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years, male or female.
2. Elective general anesthesia for surgery.
3. Operative time ≥ 30 min.
4. Preoperative body temperature within the normal range.
5. Normal preoperative bleeding and clotting time.

Exclusion Criteria:

1. Mental illness.
2. High or low basal hypothermia with high or low metabolic disease (patients with central hyperthermia include those with cerebrovascular vascular disease, traumatic brain injury and brain surgery, epilepsy, central hyperthermia due to acute hydrocephalus; thermoregulatory abnormalities including malignant hyperthermia (MHS), neuroleptic malignant syndrome and those with definite evidence of diagnosed hypo- or hyperthyroidism and current abnormal thyroid function).
3. Impaired skin insulation barriers such as large skin burns.
4. Infectious fever.
5. Other causes of body temperature above 38.5 °C three days before surgery.
6. Other persons deemed unsuitable by the investigator to participate in the clinical trial.
7. Refusal to sign the informed consent form.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1360 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative hypothermia | Up to 24 hours, from the time of entry into the operating room to the time of exit from the operating room.
  Intraoperative hypothermia, defined as a core temperature below 36 °C

SECONDARY OUTCOMES:
Postprocedural Shivering | up to 60 minutes
  A compensatory response of the body to hypothermic stimuli that cause rapid rhythmic，Once the procedure is completed, the patient will be extubated and the presence or absence of shivering will be recorded up to 60 minutes after the extubation with the Badjatia 2008 scale consisting of a gradual evaluation of 0 to 3 points. With scores greater or equal to 1, shivering is considered established. contraction of skeletal muscle for thermogenesis
Intraoperative bleeding volume | up to 24 hours after surgery
  Routine intraoperative monitoring indicators
Postoperative blood count | up to 24 hours after surgery
  The number of red blood cells, white blood cells and platelets in the blood is calculated by smearing the blood in a routine blood test and looking at it under the microscope.
30-day postoperative readmission | 30 days after surgery
  Routine postoperative monitoring indicators
6-month postoperative complications (surgical complications, pulmonary infections, blood clots) | 6 months after surgery
  Routine postoperative monitoring indicators
30-day postoperative complications (surgical complications, pulmonary infections, blood clots) | 30 days after surgery
  Routine postoperative monitoring indicators
30-day postoperative mortality | 30 days after surgery
  Routine postoperative monitoring indicators
Postoperative coagulation index | up to 24 hours after surgery
  Routine intraoperative monitoring indicators
Intraoperative blood transfusion volume | 15 minutes before the end of the surgery
  Routine intraoperative monitoring indicators, recorded according to intraoperative blood transfusion volume
Intraoperative fluid transfusion | 15 minutes before the end of the surgery
  Routine intraoperative monitoring indicators, the general rehydration amount for surgical patients is 4-6 ml per kilogram of body weight per hour
intraoperative flushing fluid volume | 15 minutes before the end of the surgery
  Routine intraoperative monitoring indicators, record the amount of intraoperative irrigation fluid used, depending on the procedure
Shivering severity | 60 minutes
  The post operative shivering scale of Badjatia 2008 will be used. It consist of a gradual evaluation of 0 to 3 points, with 0 being the absence of shivering, 1 slight shivering, 2 moderate and 3 severe. The highest score obtained will be recorded within the measurements made every 5 minutes in the first 60 minutes after extubation.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No